CLINICAL TRIAL: NCT05555212
Title: Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of QLH11811 in Advanced or Metastatic NSCLC Patients Who Have Progressed After EGFR-TKI Treatment
Brief Title: To Evaluate the Efficacy of QLH11811 in Advanced NSCLC Patients With EGFR Mutation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QLH11811
Record Dates: First submitted 2022-08-23; First posted 2022-09-26 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2022-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: This is a phase 1, open-label, dose escalation and cohort expansion study and conducted in China and the United States to investigate the safety, tolerability and preliminary efficacy of QLH11811 in advanced or metastatic NSCLC patients who have progressed after prior EGFR-TKI treatment. The study consists of the following 2 phases: phase 1: dose escalation (1a) and phase 2: cohort expansion (1b), as detailed in Overall Schematic of Study Design. Phase 1a: this dose escalation study will be conducted in China and the United States, respectively, and the dose escalation will start from starting dose in China and from dose level next to the MTD determined in Chinese subjects in the United States. Phase 1b: after the determination of RP2D, this cohort expansion study will be conducted in China and the United States concurrently to observe the safety, tolerability and efficacy of QLH11811 in advanced NSCLC patients who have EGFR mutation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dose escalation (in China) (Experimental)
  Interventions: Drug: QLH11811

INTERVENTIONS:
Drug: QLH11811 — In Ia phase, subjects will first receive oral single dose of QLH11811, then will be observed for 7 days. If the drug is tolerated by the subjects, the subjects will continue to receive the oral repeat dose of QLH11811 for 21 consecutive days. Upon the completion of observation for DLT in the subjects (DLT observation period is the 28 days after the first dose), the subjects will continue to receive the repeat dose of QLH11811 in Cycle 2 and subsequent cycles. The dosing frequency in Cycle 2 and subsequent cycles is once daily, and each cycle has 3 weeks.
  The RP2D of QLH11811 is determined on the basis of comprehensive evaluation of all safety and tolerability data and all available PK, PD and efficacy data during the dose escalation phase. In phase 1b, the cohort expansion study is carried out for all cohorts in China and the United States concurrently according to the determined RP2D.

SUMMARY:
This is a phase 1, open-label, dose escalation and cohort expansion study and conducted in China and the United States to investigate the safety, tolerability and preliminary efficacy of QLH11811 in advanced or metastatic NSCLC patients who have progressed after prior EGFR-TKI treatment. The study consists of the following 2 phases: phase 1: dose escalation (1a) and phase 2: cohort expansion (1b).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who participate voluntarily, sign informed consent form (ICF), and will be able to follow the study procedures;
2. Aged ≥ 18 years;
3. Patients who are histologically or cytologically diagnosed with EGFR mutation and have unresectable locally advanced or recurrent/metastatic NSCLC;
4. EGFR mutation requirements:

   Dose escalation phase (phase 1a): NSCLC patients who have progressed after standard EGFR-TKI treatment or cannot tolerate standard of care;

   Cohort expansion phase (phase 1b):
   1. Cohort 1: advanced NSCLC patients who have progressed after treatment with third-generation EGFR-TKIs and have EGFR C797S mutation.
   2. Cohort 2: advanced NSCLC patients who have progressed after standard EGFR-TKI treatment but have no other additional driver gene mutation(s).
   3. Cohort 3: advanced NSCLC patients who have progressed after EGFR-TKI treatment and have T790M mutation.
   4. Cohort 4: patients with locally progressed, unresectable or recurrent metastatic NSCLC who are naive to EGFR-TKI treatment and have 19del or 21L858R mutation among EGFR sensitive mutations.
5. Patients who agree to provide tumor samples (fresh tissues or archived samples) for analysis of EGFR gene.

   Dose escalation phase: tumor samples collected from the progression site of disease during or after PD after the last TKI treatment should be provided for new genetic testing The subjects who fail to provide tumor samples will be allowed to enroll only after communication and consultation with the sponsor.

   Cohort expansion phase:

   Cohort1: tumor samples collected from the progression site of disease during or after PD after the last TKI treatment should be provided for genetic testing at central laboratory.

   Cohorts 2 and 3: tumor samples collected from the progression site of disease during or after PD after the last TKI treatment should be provided for genetic testing. The genetic testing will be exempted if subjects have the test results meeting the above requirements before their enrollment.

   Cohort 4: tumor samples collected from the progression site of disease during or after PD after the last treatment should be provided for genetic testing (of EGFR mutation); and if subjects are treatment-naive, they will be required to provide the tumor samples only during the screen period. The genetic testing will be exempted if subjects have the test results meeting the above requirements before their enrollment.
6. ECOG ≤ 1 point (for details, refer to Appendix 2 ECOG performance status score);
7. Life expectancy ≥ 12 weeks;
8. Patients who have been diagnosed according to RECIST v1.1 and have measurable lesions as documented by computed tomography (CT) and/or magnetic resonance imaging (MRI) (note: subjects who do not have measurable lesions are allowed to be enrolled in phase 1a study). Note: a measurable lesion for response evaluation has to meet the following criteria: a) it is not in an area that has been involved in prior radiotherapy, or b) there is notable radiographic evidence of progression after the completion of radiotherapy and before study enrollment;
9. Patients who have adequate organ functions and meet the following criteria:

   1. Hematology:

      Absolute neutrophil count ≥ 1.5 × 109/L; platelet count ≥ 100 × 109/L; hemoglobin ≥ 90 g/L (no blood transfusion and no use of granulocyte colony stimulating factor in the 14 days prior to the screening);
   2. Coagulation:

      For patients who have not received anticoagulant therapy: international normalized ratio (INR) of prothrombin time and partial thromboplastin time ≤ 1.5 × ULN;
   3. Liver:

      Alanine aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 3.0 × ULN. For patients with liver metastases: ALT and AST ≤ 5 × ULN, total bilirubin ≤ 1.5 × ULN. For patients with Gilbert syndrome: conjugated bilirubin within normal range;
   4. Kidney:

   Serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min (calculated according to Cockcroft-Gault formula, refer to Appendix 4 Creatinine clearance calculation formula).
10. All acute toxic reactions arising from prior antineoplastic therapy or surgery have resolved to baseline or reduced in severity to ≤ Grade 1 according to NCI CTCAE V5.0 (except for alopecia or other toxicities which, in the opinion of the investigator, pose no safety risk to the patient);
11. Patients (both female and male) who agree to take effective contraceptive measures from their signing of ICF to 6 months after the last dose of the study drug. For women of childbearing potential: negative serum pregnancy test result in 7 days prior to the start of treatment is required.

Exclusion Criteria:

1. Patients who have received systemic anticancer therapies (e.g., chemotherapy, molecularly targeted therapy, radiotherapy, biotherapy, hormone therapy, vaccine therapy), or antineoplastic TCM therapy in the 2 weeks prior to the first dose of study treatment; or who have received immune-checkpoint inhibitor therapy in the 4 weeks prior to the first dose of study treatment;
2. Patients who have received radical radiotherapy (including radiotherapy of more than 25% of bone marrow) in the 4 weeks prior to the first dose, or who have received local palliative radiotherapy for bone metastatic lesions in the 1 week prior to the first dose;
3. Patients who have received strong or moderate CYP3A, P-gp inhibitors in the 1 week prior to the first dose or in 5 half-lives of these drugs (whichever is longer), or need to continue to receive these drugs during the study; and who have received strong or moderate CYP2B6, CYP1A2 and CYP3A inducers in the 4 weeks prior to the first dose;
4. Patients who are in the treatment period of other interventional clinical studies in the 4 weeks prior to the first dose. However, participants of non-interventional clinical studies (e.g., epidemiologic studies) are eligible for enrollment in this study. Patients in the survival follow-up period of interventional clinical studies are also eligible for enrollment in this study;
5. Patients who have active bacterial, fungal or viral infection requiring systemic therapies within the 1 week prior to the first dose;
6. Patients who have underwent a major operation (e.g., a surgical operation requiring local or general anesthesia and hospitalization) in the 3 weeks prior to the start of study treatment;
7. Patients with a history of chronic diarrhea, including but not limited to Crohn's disease, irritable bowel syndrome, etc.;
8. Patients who have experienced > CTCAE Grade 1 continuous diarrhea within the 1 week prior to the first dose;
9. Patients with serious respiratory disorders, e.g. interstitial lung disease, radiation pneumonitis, drug-induced pneumonia (however, patients whose conditions have resolved and stabilized for 3 months or more are eligible for enrollment);
10. Patients with symptomatic metastasis to central nervous system (CNS) and/or with meningitis carcinomatosa.

    Note: patients with brain metastases whose clinical symptoms have stabilized after treatment are eligible for participation in the study, provided that their conditions are radiographically stabilized (defined as stability demonstrated by 2 brain images acquired by the same imaging technique after treatment of brain metastases). These imaging scans should be carried out at an interval of at least 4 weeks, and show no signs of intracranial progression. Furthermore, brain metastases or its treatment induced neurologic symptoms need to regress to baseline level or resolve. All steroids administered as a part of the treatment must be completed ≥ 3 days prior to the administration of study treatment.
11. Patients with clinically significant cardiovascular and cerebrovascular diseases, including but not limited to:

    1. Myocardial infarction or unstable angina in the 6 months prior to the first dose;
    2. Stroke or transient ischemic attack in the 6 months prior to the first dose;
    3. Any clinically significant abnormalities in resting ECG in terms of cardiac rhythm, heart rate, conduction or morphology, e.g. complete left bundle branch block, third-degree conduction block, second-degree conduction block, PR interval > 250 ms, etc.;
    4. Uncontrolled hypertension after active treatment: systolic pressure > 180 mmHg or diastolic pressure > 100 mmHg;
    5. Congestive cardiac failure (NYHA functional class III-IV);
    6. Pericarditis or clinically significant pericardial effusion;
    7. Myocarditis;
    8. 12-lead ECG shows that mean QT interval (QTcF) > 450 ms (male) or > 470 ms (female) before the first dose of investigational drug;
    9. Failure to discontinue the drugs that may cause QTc prolongation or torsades de pointes (e.g., antiarrhythmics) during the study.
12. Patients with clinically uncontrolled serous effusion(e.g., pleural fluid that cannot be controlled by drainage or other methods).
13. Patients with active gastrointestinal disorders or other conditions that have serious interference with the drug absorption.
14. Patients with any condition that have an adverse impact on the swallowing of the drug or on the absorption or PK parameters of the investigational drug;
15. Patients with known serious allergy to the study drug or any excipient of the drug;
16. Patients with known HIV test positive result and/or treponema pallidum antibody test positive result (except for those whose infection has been cured after treatment).
17. Patients with HBsAg positive result and HBV DNA > 2000 IU/mL or 104 copies/mL (for sites which only provide the qualitative testing, HBV DNA test result is positive or higher than lower limit of detection); or with HCV antibody positive and HCV RNA positive results.
18. Patients who experienced other malignancies (with the exceptions of Bowen's disease; cured basal cell or squamous cell skin cancer; prostate cancer with a Gleason score of 6; treated cervical carcinoma in situ) in the 2 years prior to the study enrollment.
19. Pregnant or lactating women. Lactating female subjects need to stop breast-feeding before the first dose of study treatment, which cannot be resumed throughout the study and in the 6 months after the last dose of study treatment.
20. Patients with any existing serious or unstable diseases (except for the above-mentioned malignancies), psychiatric disorders or any disease or medical condition which, in the investigator's opinion, may have an adverse impact on the subject safety, the signing of ICF or the compliance with the study procedures.
21. Patients who are currently participating in a clinical study of other investigational therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety parameters | 2 years
  adverse events (AEs), serious adverse events (SAEs) and other safety results
ORR | 2 years
  Objective response rate (ORR) (evaluated by the Independent Review Committee in NSCLC patients who have EGFR-C797S mutation according to RECIST v1.1).

SECONDARY OUTCOMES:
Possible metabolites of QLH11811 in plasma | 6 month
  QLH11811 metabolites that may be present in the blood were detected

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Pharmaceutical.Co.,Ltd, Jinan, Shandong, China